CLINICAL TRIAL: NCT05076851
Title: A Randomized, Controlled, Double-blind, Single Center，Clinical Trial to Evaluate the Efficacy and Safety of Neoadjuvant Therapy With Proxalutamide Combined With Androgen Deprivation Therapy（ADT）for High Risk Prostate Cancer
Brief Title: Neoadjuvant Therapy With Proxalutamide Combined With Androgen Deprivation Therapy（ADT）for High Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongqian Guo (Other)
Responsible Party: Sponsor-Investigator, Hongqian Guo, chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-GT0918-CN-1008
Record Dates: First submitted 2021-06-22; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Neoadjuvant Therapy \High Risk Prostate Cancer
MeSH Terms: interventions — proxalutamide

STUDY DESIGN:
Intervention Model Description: Proxalutamide: androgen deprivation therapy（ADT）=2:1
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): placebo+ADT
  Interventions: Other: placebo
- Proxalutamide (Experimental): Proxalutamide +ADT
  Interventions: Drug: Proxalutamide

INTERVENTIONS:
Other: placebo — placebo+ADT（Androgen Deprivation Therapy） ，Route of placebo administration: tablet, dosage：300mg , dosage form oral , frequency of administration：QD
  Arms: placebo group
Drug: Proxalutamide — Proxalutamide +ADT（Androgen Deprivation Therapy） ，Route of Proxalutamide administration: tablet, dosage：300mg , dosage form oral , frequency of administration：QD
  Arms: Proxalutamide

SUMMARY:
This trial aims to evaluate the efficacy and safety of neoadjuvant therapy with Proxalutamide combined with androgen deprivation therapy（ADT）for High risk prostate cancer ，This trial is A randomized, controlled, double-blind, single center.Treatment cycle is 6 months,

ELIGIBILITY:
Inclusion Criteria:

1. Patients must participate voluntarily and sign an informed consent form (ICF), indicating that they understand the purpose and required procedures of the study
2. Patients must be ≥ 18，male
3. Histopathological by Prostate biopsy confirmed prostatic cancer（No Neuroendocrine prostate cancer or small cell carcinoma）
4. High-risk prostate cancer (T2c≤ clinical stage ≤T4 or Gleason score ≥8 or PSA≥20ng/ml)
5. Patients willing to undergo laparoscopic radical resection of prostate cancer and extensive lymph node dissection
6. ECOG PS：0-1

Exclusion Criteria:

1. Imaging or biopsy confirmed distant Metastatic lesion
2. The number of regional lymph nodes metastasis >3
3. Patients had undergone The treatment of Systemic chemotherapy and endocrine therapy for prostate cancer
4. Patients had undergone prostate surgery、radical radiotherapy or Bilateral orchidectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | up to 6months
  The proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy
Proportion of Subjects With Minimal Residual Disease | up to 6months
  The proportion of subjects that have residual tumors with maximum diameter of 3 mm or less after radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Phd, Study Chair — Study Chair Department of Urology, Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China